CLINICAL TRIAL: NCT07087249
Title: Efficacy of Ultrasound Biofeedback in Brazilian Childhood Apraxia of Speech: A Randomized Clinical Trial
Brief Title: Efficacy of Ultrasound Biofeedback in Brazilian Childhood Apraxia of Speech
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aline Mara de Oliveira (Other)
Responsible Party: Sponsor-Investigator, Aline Mara de Oliveira, Principal Investigator, Santa Catarina Federal University
Organization: Santa Catarina Federal University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09476918.5.0000.0121
Record Dates: First submitted 2025-07-06; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Childhood Apraxia of Speech; Speech Sound Disorders
Keywords: Speech Therapy; Motor Speech Disorder; Childhood Apraxia of Speech; Verbal Dyspraxia; Ultrasound Biofeedback
MeSH Terms: conditions — Apraxias; Speech Sound Disorder; Communication Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel arms: (1) experimental group with ultrasound visual biofeedback; (2) control group with traditional speech therapy.
Who Masked: Outcomes Assessor
Masking Description: Only the person assessing post-treatment outcomes will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: Ultrasound Visual Feedback (Experimental): Speech therapy using real-time ultrasound imaging to provide visual feedback of tongue movement. Designed for children with Childhood Apraxia of Speech (CAS). Sessions occur twice per week for six weeks (12 total), targeting speech motor planning and accuracy using motor learning principles.
  Interventions: Behavioral: Ultrasound Visual Feedback
- Behavioral: Traditional Speech Therapy (Active Comparator): Speech therapy for children with Childhood Apraxia of Speech (CAS), based on motor learning principles. Sessions are delivered twice per week over six weeks (12 total).
  Interventions: Behavioral: Traditional Speech Therapy

INTERVENTIONS:
Behavioral: Ultrasound Visual Feedback — Speech therapy using real-time ultrasound imaging to provide visual feedback on tongue placement and movement. Aimed at improving speech accuracy and motor planning in children with Childhood Apraxia of Speech (CAS). The intervention follows principles of motor learning and includes 12 individual sessions over 6 weeks (twice per week). Practice alternates between ultrasound-assisted and non-assisted phases to promote generalization.
  Arms: Behavioral: Ultrasound Visual Feedback
Behavioral: Traditional Speech Therapy — Standard speech motor therapy for children with Childhood Apraxia of Speech (CAS), based on evidence-based motor learning approaches. No visual feedback tools are used. Therapy focuses on blocked and random practice, varied feedback, and increasing speech complexity. Delivered in 12 sessions over 6 weeks (twice per week).
  Arms: Behavioral: Traditional Speech Therapy

SUMMARY:
This study is a single-blind, randomized controlled trial evaluating the efficacy of ultrasound visual biofeedback (UVB) in the treatment of Childhood Apraxia of Speech (CAS) among Brazilian children. Approximately half of the participants are randomly assigned to an Experimental group receiving the ultrasound biofeedback intervention, and the other half to a Control group receiving conventional motor-based therapy without ultrasound. Randomization is performed using a computer-generated sequence (allocation ratio 1:1), with allocation concealment (e.g. sealed opaque envelopes) to prevent selection bias. Blinding is maintained for outcome assessment: an independent speech-language pathologist who is masked to group assignment will evaluate pre- and post-therapy speech samples for all children. Neither the therapists nor the participants are blinded (due to the nature of the intervention), but the use of blinded outcome evaluators helps ensure objective assessment.

DETAILED DESCRIPTION:
Ultrasound Biofeedback Intervention (Experimental Group): The experimental intervention involves intensive speech therapy augmented with real-time ultrasound tongue imaging as visual feedback. A portable ultrasound system with a small microconvex transducer is used, positioned submentally (under the child's chin) to capture a midsagittal view of the tongue.

. The ultrasound transducer emits safe, high-frequency sound waves, and the reflected signals produce a dynamic image of the tongue's surface on a monitor. Specialized software (such as Articulate Assistant Advanced (AAA) by Articulate Instruments Ltd.) is utilized to display and synchronize the ultrasound images with speech output.

During therapy, the child can see a real-time outline of their tongue moving on the screen as they attempt target sounds. This visual biofeedback serves as knowledge of performance - it allows the child to compare their tongue shape and placement against the therapist's model or a predetermined target shape. For example, the clinician may instruct the child to "lift the back of your tongue" for a velar sound and the ultrasound image immediately shows whether the child's tongue dorsum is reaching the correct position. A custom head-stabilization apparatus is often used to keep the probe steady and ensure consistent imaging. Throughout the ultrasound-assisted practice, the therapist provides cues and coaching based on the visual information (e.g. telling the child to aim the tongue toward a certain position on the screen) in addition to the typical auditory and tactile cues.

Control Intervention (Conventional Motor-Based Therapy): The control group receives an intensive motor-based speech therapy program of equal dose and duration, but without ultrasound visual feedback. This conventional therapy is grounded in established motor learning principles for CAS, focusing on repetitive practice of speech targets with gradually increasing difficulty and strategic feedback. Children in the control group practice the same type of target sounds and words as the experimental group (described below under "Therapy Targets and Sessions"). The key difference is that the clinician uses standard cueing techniques instead of instrumented biofeedback: for example, verbal descriptions of tongue placement ("Put your tongue tip behind your teeth for /t/"), visual cues (watching the clinician's mouth, using a mirror), tactile prompts, and knowledge of results feedback (indicating whether the attempt was correct or not). Both groups therefore receive high-intensity, drill-based practice and employ principles of motor learning (such as frequent practice, feedback, and gradually reduced cueing), but the experimental group gains extra visual feedback about tongue movements, whereas the control relies on traditional auditory-proprioceptive feedback only. This distinction reflects different motor learning approaches: the ultrasound provides immediate internal feedback on articulator movement, while the control approach emphasizes outcomes (sound correctness) without direct internal visual feedback.

Therapy Targets and Session Structure: Therapy targets are individualized for each child based on their speech error profile, focusing on phonemes and word shapes that are challenging due to CAS. Targets include specific phonemes (speech sounds) and various syllable structures (e.g., CV syllables, CVC words, consonant clusters, and multisyllabic words) that the child has difficulty producing. For instance, a child who cannot accurately produce lingual consonants might have targets like /s/, /ʃ/, or /k/ in simple syllables ("sa", "ka") and in words of increasing complexity ("sapato", "cavalo", etc.). Both groups practice a similar set of target stimuli (words or pseudowords containing these phonemes in different syllabic contexts), chosen to facilitate motor planning and to allow measurement of generalization to unpracticed words. Each participant undergoes a series of therapy sessions over the course of the intervention. Sessions are typically scheduled multiple times per week (e.g. 2 sessions per week) for several weeks, to accumulate a high dose of practice trials. Each session lasts about 45-60 minutes, structured into two phases: an ultrasound-assisted phase and an unassisted phase. In the experimental group's sessions, roughly the first half of the session is the ultrasound-assisted practice. During this phase (approximately 20-30 minutes), the child practices the target sounds/words while viewing the real-time ultrasound display of their tongue. The clinician might use 8-10 target words per session, training each multiple times. The child is encouraged to adjust their articulations by watching the tongue image (for example, ensuring the tongue shape reaches a certain height or contact for a sound) and by following the clinician's live feedback on the screen. In the second half of the session, the ultrasound machine is turned off (or the screen is hidden) for the unassisted practice phase, which also lasts about 20-30 minutes.

In this phase, the child continues to practice the same target words without visual feedback, relying on what they learned and on the therapist's verbal feedback. This approach - practicing first with visual guidance and then without - is designed to promote generalization of the skill beyond the immediate feedback condition. It allows the child to attempt the targets as independently as possible, simulating real speaking conditions. The therapist provides knowledge of results (indicating correct vs. incorrect productions) and faded cues as needed during the unassisted phase. The session structure is thus consistent between groups in terms of time and practice, with the experimental group's first portion using ultrasound and the control group's first portion using equivalent additional exercises without ultrasound (such as extra drilling or auditory bombardment). By the end of each session, both groups have spent equal time practicing target pronunciations; the experimental group has spent part of that time with visual biofeedback and the control group with traditional methods. Over the entire treatment course, children may receive on the order of 10-16 therapy sessions (depending on the study protocol), which is a dosage chosen based on prior CAS intervention studies. All sessions are conducted by speech-language pathologists trained in the respective therapy techniques. Parents are not present during the actual practice to avoid distractions (unless required for child compliance), but they may receive periodic updates or training on how to support practice at home (though home practice is not formally measured in this trial).

Outcome Measures and Evaluation Therapeutic efficacy is assessed by comparing pre- and post-intervention speech performance using quantitative speech measures and functional ratings. Baseline assessments include a detailed speech evaluation and a hearing screening. All children undergo a hearing screening (pure-tone audiometry or otoacoustic emissions, as appropriate for age) to confirm normal hearing ability, since uncorrected hearing loss could affect speech development. The primary speech outcome measure is the Percentage of Consonants Correct (PCC) - a standard metric of speech accuracy. To calculate PCC, children's speech is elicited through standardized tasks (such as naming pictures or repeating words/sentences), and audio recordings are phonetically transcribed by trained examiners. PCC is computed as the proportion of consonant sounds produced correctly out of the total attempted, and is expressed as a percentage. An improvement in PCC from pre- to post-therapy indicates gains in articulatory accuracy. In addition to overall PCC, consonant accuracy on treated versus untreated (generalization) words may be analyzed to see if skills carry over to new vocabulary. Speech intelligibility is another key outcome. Intelligibility refers to how well a child's speech is understood by listeners. It is evaluated using established tools such as intelligibility rating scales or parent questionnaires. For example, an independent listener or a panel of judges might rate the child's speech on a scale (e.g., 1 = mostly unintelligible, 5 = completely intelligible) or classify each test word as understandable or not. Alternatively, the Intelligibility in Context Scale (ICS) (a parent-reported measure) could be used to gauge improvements in everyday communication. By assessing intelligibility before and after treatment, the study can determine if the child's functional communication has improved, not just their articulation of individual sounds. Secondary outcome measures may include speech consistency and motor planning skills (for instance, measuring changes in the variability of repeated attempts, or using a tool like the Dynamic Evaluation of Motor Speech Skill for diagnostic confirmation), as well as prosody (the rhythm and stress of speech), since CAS often affects stress patterns. If applicable, the trial will examine whether the ultrasound biofeedback has any added benefit for prosodic accuracy or consistency of speech movements compared to the control therapy. All post-treatment outcome assessments are conducted by evaluators who are blinded to group allocation and to the time point of the sample (pre- vs. post-therapy). Typically, the pre- and post-therapy speech samples are recorded and randomized so that the blinded evaluators cannot tell which is which. They then perform the transcription and ratings without knowing whether a given sample is from before or after treatment, or whether the child was in the experimental or control group. This blinding minimizes bias in scoring. In summary, this trial provides a thorough examination of an ultrasound-based intervention for CAS. The experimental UVB protocol is detailed with specific equipment (ultrasound machine, transducer, and software) and a clearly defined visual feedback mechanism. The evaluation framework employs objective measures like PCC and intelligibility scales to capture changes in speech production, all under rigorous conditions of randomization and blinded assessment. The experimental group and control group interventions are carefully matched in structure and grounded in motor learning principles, differing primarily in the presence or absence of real-time ultrasound tongue imaging. This design will allow us to determine whether ultrasound visual feedback offers a significant advantage in improving the speech of children with CAS, beyond what can be achieved with traditional therapy alone.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Childhood Apraxia of Speech (CAS) confirmed by at least two certified speech-language pathologists; Aged between 5 and 16 years; Monolingual Brazilian Portuguese speakers; Normal hearing, cognitive, and receptive language skills; Normal results on oral-facial and non-verbal intelligence screenings.

Exclusion Criteria:

Hearing impairment or auditory processing disorders Neurological, intellectual, or anatomical conditions affecting speech (e.g., cleft palate, cerebral palsy, dysarthria) Diagnosis of global motor developmental disorders Bilingual speakers or those exposed to other languages at home

Ages: 5 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-08-06 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Correct Consonants (PCC) | Assessed at follow-up, 4 weeks after final therapy session.
  Percentage of correctly produced consonants(PCC) for treated and untreated stimuli: Generalization to novel words, phrases, sentence contexts and spontaneous speech; Maintenance of gains at follow-up;

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Aline Mara de Oliveira, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to ethical and privacy considerations in accordance with Brazilian data protection laws and institutional review board policies.

REFERENCES:
- [Background] Cleland J, McCluskey R, Dokovova M, Crampin L, Campbell L. A mixed-methods pilot randomized control trial of ultrasound visual biofeedback versus standard intervention for children with cleft palate +/- cleft lip: Parents' and children's perspectives. Int J Lang Commun Disord. 2025 Jan-Feb;60(1):e13144. doi: 10.1111/1460-6984.13144. PMID 39651790
- [Background] McCabe P, Preston JL, Evans P, Heard R. A Pilot Randomized Control Trial of Motor-Based Treatments for Childhood Apraxia of Speech: Rapid Syllable Transition Treatment and Ultrasound Biofeedback. Am J Speech Lang Pathol. 2023 Mar 9;32(2):629-644. doi: 10.1044/2022_AJSLP-22-00144. Epub 2023 Feb 27. PMID 36848673